CLINICAL TRIAL: NCT00261313
Title: An Open Label Phase 2 Study of Doxorubicin and Cyclophosphamide Followed by Paclitaxel Delivered Every 14 Days With Pegfilgrastim and Darbepoetin Alfa Support for the Adjuvant Treatment of Women With Breast Cancer
Brief Title: ACCELERATE: Doxorubicin and Cyclophosphamide Followed by Paclitaxel With Pegfilgrastim and Darbepoetin Alfa Support for the Treatment of Women With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040137
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Doses dense chemotherapy; Growth factor support; Adjuvant Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pegfilgrastim; Darbepoetin alfa

ARMS (2):
- Aranesp (Experimental)
  Interventions: Drug: Aranesp
- Neulasta (Experimental)
  Interventions: Drug: Neulasta

INTERVENTIONS:
Drug: Neulasta — 6mg Neulasta to be given approximately 24 hours afer each cycle of chemotherapy
  Arms: Neulasta
Drug: Aranesp — If Hb drops below 110, 300mcg Aranesp will be administered.
  Arms: Aranesp

SUMMARY:
This is a study of dose dense doxorubicin/cyclophosphamide (AC) followed by paclitaxel (Taxol; T) with pegfilgrastim (Neulasta) and darbepoetin alfa support in the adjuvant breast cancer setting.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis node-positive or high risk node negative
* Estrogen receptor (ER) negative or ER positive (stage IIA, IIB or IIIA) disease.

Exclusion Criteria:

* Metastatic breast cancer
* Clinically significant cardiac disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-12; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects experiencing any delay in any cycle of chemotherapy over the course of the study | 3 months

SECONDARY OUTCOMES:
Febrile neutropenic events and adverse event profile will be assessed | 4 months
To assess chemotherapy and subject dose delays and reductions which are specific and/or non specific to haematological toxicities | 3 months
Frequency of red blood cell (RBC) transfusions | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com